CLINICAL TRIAL: NCT02543333
Title: Validation of Structured Light Plethysmography: Pre- and Post- Bronchodilator Challenge
Brief Title: Validation of Structured Light Plethysmography: Asthma
Acronym: SLPBD
Status: Completed | Type: Observational
Sponsor: Pneumacare Ltd (Industry)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); University Hospitals of North Midlands NHS Trust (Other); Keele University (Other)
Responsible Party: Sponsor
Other Study IDs: PMC-T3D-002/2
Record Dates: First submitted 2015-08-28; First posted 2015-09-07 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Asthma
Keywords: Acute Asthma,
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Asthma: Patients attending outpatient clinic as part of their clinical care who have FEV1 less than 80% of predicted and are referred by their clinician for a bronchodilator test
- Acute Asthma: Inpatients admitted for an acute asthma exacerbation
- Normal: Participants with no current or previous diagnosis of a respiratory condition

SUMMARY:
Validation of Structured Light Plethysmography (SLP) in patients with asthma, in patients with acute asthma; an observational study in healthy participants and during patients' clinical investigation of broncho-reversibility in the asthma groups.

DETAILED DESCRIPTION:
A non-randomised observational study to validate Structured Light Plethysmography in three groups of participants: those with stable asthma and those with acute asthma, who are undergoing routine clinical investigation of broncho-reversibility using spirometry. We will also observe a normal healthy group who will receive no clinical intervention. SLP data capture and spirometry (as part of the patients clinical care) will be performed before and after a Bronchodilator reversibility test which is part of the patients normal clinical care (except in the normal healthy group where no bronchodilator will be given). The data collected from this study will allow us to examine the effect of bronchodilators on breathing patterns in these patients and also compare breathing patterns in asthma patients to those in healthy individuals.

The participant will wear a plain white t-shirt. Alternatively, the measurement can be taken on bare skin or with the participant (if female) wearing a plain material white bra. The participant is asked to sit down on a chair or lie down with their neck in a neutral position and their back as straight as possible in front of the SLP device (Thora-3Di, Pneumacare Ltd). The projector is lined up to project the grid of light over the participant's chest and upper abdomen. and will be instructed to perform a period of 5 minutes of tidal breathing, They will otherwise be asked to remain as still as possible throughout the measurement. During the sequence of breathing, thoracoabdominal wall movements will be captured by the device.

participant on completion of their Bronchodilator Challenge within the Lung Function Department or clinic

The SLP measurement is repeated on completion of their Bronchodilator reversibility test within the Lung Function Department or clinic.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 2 and 80 years

Exclusion Criteria:

* Patients with significant co morbidities resulting in clinical instability (assessed by the clinician at screening only):
* obstructive sleep apnea, Apnoea hypopnoea index > 30 (if known)
* An acute or chronic condition that, in the investigator's opinion, would limit the patient's ability to participate in the study
* BMI > 40
* Inability to consent/comply with trial protocol

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 100 participants between the ages of 2 and 80 with stable asthma who are undergoing routine clinical investigation of broncho-reversibilty.
  100 participants between the ages of 2 and 80 with acute asthma who are undergoing routine clinical investigation of broncho-reversibilty.
  100 participants between the ages of 2 and 80 with no history of respiratory disease ('Normal'). These participants will not undergo a bronchodilator challenge.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in SLP Parameters after Bronchodilator Reversibility Test | Baseline and 15 minutes after bronchodilator reversibility test (in asthma patients)
  SLP breathing parameters derived from the movement of the thoracoabdominal (TA) wall during tidal breathing.
Difference in SLP Parameters between Asthma Patients and Healthy Subjects | Baseline
  SLP breathing parameters derived from the movement of the thoracoabdominal (TA) wall during tidal breathing.

SECONDARY OUTCOMES:
Change from Baseline in Forced Expiratory Volume in 1 second (FEV1) after Bronchodilator Reversibility Test | Baseline and 15 minutes after bronchodilator reversibility test (in asthma patients)
  Measurement of FEV1 before and after bronchodilator
Change from Baseline in Forced Vital Capacity (FVC) after Bronchodilator Reversibility Test | Baseline and 15 minutes after bronchodilator reversibility test (in asthma patients)
  Measurement of FEV1 before and after bronchodilator

CONTACTS AND LOCATIONS:
Overall Officials: Richard Iles, MD, Principal Investigator — Cambridge University Hospitals Trust
Locations (2):
- United Kingdom (2):
  - Cambridge University Hospitals Foundation Trust, Cambridge, Cambridgeshire
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire

REFERENCES:
- [Background] Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. General considerations for lung function testing. Eur Respir J. 2005 Jul;26(1):153-61. doi: 10.1183/09031936.05.00034505. No abstract available. PMID 15994402
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] de Boer WH, Lasenby J, Cameron J, Wareham R, Ahmad S, Roach C, Hills W, Iles R. SLP: a zero-contact non-invasive method for pulmonary function testing. In: Labrosse F, Zwiggelaar R, Liu Y, Tiddeman B, eds, Proceedings of the British Machine Vision Conference. BMVA Press, 2010; pp 85.1-85.12
- [Background] Morgan MD, Gourlay AR, Denison DM. An optical method of studying the shape and movement of the chest wall in recumbent patients. Thorax. 1984 Feb;39(2):101-6. doi: 10.1136/thx.39.2.101. PMID 6701820
- [Derived] Hmeidi H, Motamedi-Fakhr S, Chadwick EK, Gilchrist FJ, Lenney W, Iles R, Wilson RC, Alexander J. Tidal breathing parameters measured by structured light plethysmography in children aged 2-12 years recovering from acute asthma/wheeze compared with healthy children. Physiol Rep. 2018 Jun;6(12):e13752. doi: 10.14814/phy2.13752. PMID 29932498